CLINICAL TRIAL: NCT00020488
Title: A Phase I & Pharmacologic Trial Of Sequential Irinotecan As A 24-Hour IV Infusion, Leucovorin, & Flurouracil As A 48-Hour IV Infusion In Adult Cancer Patients
Brief Title: Combination Chemotherapy in Treating Patients Who Have Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068548; NCI-01-C-0082; MB-NAVY-00-02; MB-NAVY-B00-038; NCT00021515 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2003-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended phase II dose of irinotecan, leucovorin calcium, and fluorouracil in patients with advanced solid tumors.
* Determine the toxic effects of this regimen in these patients.
* Determine the pharmacokinetic and pharmacodynamic profiles of irinotecan and fluorouracil in patients treated with this regimen.
* Determine the correlation of polymorphisms in the promoter region of the thymidylate synthase gene with clinical toxicity and response in patients treated with this regimen.
* Determine the correlation of polymorphisms in the uridine diphosphate glucuronosyltransferase 1A1 gene promoter with the extent of SN-38 glucuronidation and severity of diarrhea in patients treated with this regimen.
* Assess any anti-tumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of irinotecan and fluorouracil.

Patients receive irinotecan IV continuously over 24 hours on days 1 and 15 and leucovorin calcium IV over 30 minutes followed by fluorouracil IV continuously over 48 hours on days 2 and 16. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. Once the MTD of irinotecan has been determined, additional cohorts receive escalating doses of fluorouracil until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor that has failed standard therapy or for which no standard therapy exists

  * Locally advanced, unresectable, primary or recurrent disease OR
  * Metastatic disease
* Previously untreated disease allowed provided this regimen represents reasonable first-line therapy
* No leukemia or lymphoma
* No primary CNS malignancy or CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.6 mg/dL
* AST/ALT no greater than 4 times upper limit of normal

Renal:

* Creatinine no greater than 1.6 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other serious concurrent illness that would preclude study
* No active infection requiring IV antibiotics
* No known hypersensitivity to irinotecan
* No marked intolerance to fluorouracil

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* More than 4 weeks since prior chemotherapy (at least 6 weeks for nitrosoureas or mitomycin) and recovered
* Prior short-infusion irinotecan allowed
* Prior fluorouracil allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 2 weeks since prior radiotherapy and recovered
* At least 8 weeks since prior strontium chloride Sr 89

Surgery:

* Recovered from prior surgery

Other:

* No concurrent cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szabo, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States